CLINICAL TRIAL: NCT05138159
Title: A Prospective, Phase II, Single-arm Study to Evaluate The Safety and Efficacy of Donafenib Plus S-1 in Treating Patients With Metastatic Pancreatic Cancer After Chemotherapy With Nab-paclitaxel Plus Gemcitabine Regimen
Brief Title: A Study of Donafenib Plus S-1 in Treating Patients With Metastatic Pancreatic Cancer After Chemotherapy With Nab-paclitaxel Plus Gemcitabine Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDAC-ZPS-S
Record Dates: First submitted 2021-11-17; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — donafenib; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Donafenib + S-1 (Experimental): Donafenib: 200mg po bid； S-1 capsule: According to the body surface area <1.25m2 40mg/d, 1.25 ~ 1.5 m2 50 mg/d, > 1.5m2 60mg/d po bid, taking 14 days, stopping for 7 days, 21 days for 1 cycle.
  Interventions: Drug: Donafenib; Drug: S1

INTERVENTIONS:
Drug: Donafenib — Donafenib: 200mg po bid.
Drug: S1 — S-1 capsule: According to the body surface area <1.25m2 40mg/d, 1.25 ~ 1.5 m2 50 mg/d, > 1.5m2 60mg/d po bid, taking 14 days, stopping for 7 days, 21 days for 1 cycle.

SUMMARY:
This is a single arm, open label Phase II clinical trial to evaluate the efficacy and safety of donafenib combined with S-1 in treating Patients with metastatic pancreatic cancer after chemotherapy with Nab-paclitaxel plus gemcitabine regimen.

DETAILED DESCRIPTION:
While NG ( Nab-paclitaxel + gemcitabine) is one of the preferred first-line chemotherapy for metastatic pancreatic cancer, we have to investigate possible therapeutic options after NG regimen. In this single arm, open-label clinical trial, metastatic pancreatic cancer patients will be received donafenib and S-1. Treatment repeats every 3 weeks until the disease recurrence or unacceptable toxicity, death or begin a novel therapeutic.

The efficacy and safety data will be assessed through OS, ORR, DCR, PFS,TTP and adverse effects as graded by NCI CTC-AE 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and willing to complete the study according to the protocol.
* Age ≥ 18 years and ≤ 75 years, and there is no limit on the gender
* ECOG performance scale 0-1;
* Diagnosed as pancreatic adenocarcinoma by histology and cytology;
* Treatment of patients with advanced metastatic pancreatic cancer who have failed with NG (Nab-paclitaxel + gemcitabine) regimen(The disease progresses during the course of treatment or within 6 months after the end of treatment, with clear imaging evidence; this does not include patients with intolerable toxicity)；
* Baseline blood routine and biochemical indexes meet the following criteria:

  1. Blood routine examination criteria must be met: (no blood transfusion within 14 days)

     1. HB≥90g/L；
     2. ANC≥1.5×109/L；
     3. PLT≥100×109/L.
  2. Biochemical tests are subject to the following criteria:

     1. BIL <1.25xULN ；
     2. ALT and AST<2.5ULN；
     3. Serum creatinine. Less than 1.5 times the upper limit of normal value, Endogenous creatinine clearance>60ml/min ( Cockcroft-Gault formula).
     4. Albumin≥28g/L.
  3. Blood coagulation indexes are subject to the following criteria:

     1. Prothrombin time (PT) and international normalized ratio (INR) ≤1.5 × ULN;
     2. Activated partial thromboplastin time（APTT）≤1.5 × ULN.
* According to the standard of RECIST 1.1, there is at least one imaging measurable lesion;
* Life expectancy ≥ 3 months;
* Patients and their families were willing to cooperate with follow-up.

Exclusion Criteria:

* Diagnosis of malignant diseases other than pancreatic cancer within 5 years prior to first administration (excluding cured skin basal cell carcinoma, squamous carcinoma of the skin, and/or resected carcinoma in situ);
* Medical conditions that affect absorption, distribution, metabolism, or clearance of the study drug (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorders, etc.);
* Patients with brain metastases or pial metastases;
* Patients with a clear past history of neurological or psychiatric disorders, including epilepsy or dementia;
* Comorbidities (e.g., severe or uncontrolled hypertension, severe diabetes, and/or thyroid disease) that, in the investigator's judgment, seriously endanger patients' safety or prevent them from completing the study;
* The patient was currently participating in an interventional clinical study or had been treated with another study drug or study device in the 4 weeks prior to initial dosing;
* The patient had a history of organ transplantation;
* Concurrent administration of drugs that may prolong QTc and/or induce Tdp;
* Patients also take drugs that affect drug metabolism;
* HIV infection or acute or chronic viral hepatitis (hbSAG positive, HBV-DNA load ≥500IU/ml and/or HCV antibody positive);
* Excluded patients with serious cardiovascular disease, including grade ≥II cardiac dysfunction (NYHA criteria);
* Patients with severe gastrointestinal dysfunction (bleeding, infection, obstruction, or diarrhea greater than grade 1) were excluded;
* Patients with abnormal coagulation function, bleeding tendency, or receiving thrombolytic or anticoagulant therapy were excluded;
* Patients with a severe arterial thromboembolism event within 6 months were excluded;
* Excluding women who are pregnant or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | through study completion, an average of 1 year
  To evaluate the overall survival of patients with advanced metastatic pancreatic cancer who have failed with NG (Nab-paclitaxel + gemcitabine) regimen after treatment with Donafenib combined with S-1.

SECONDARY OUTCOMES:
Progression Free Survival | through study completion, an average of 1 year
  To investigate the progression-free survival (PFS) of patients with advanced metastatic pancreatic cancer who have failed with NG (Nab-paclitaxel + gemcitabine) regimen after treatment with Donafenib combined with S-1.
Overall Response Rate | through study completion, an average of 1 year
  To evaluate the overall response rate of patients with advanced metastatic pancreatic cancer who have failed with NG (Nab-paclitaxel + gemcitabine) regimen after treatment with Donafenib combined with S-1.
Incidence of Adverse Events | through study completion, an average of 1 year
  Adverse events of patients with advanced metastatic pancreatic cancer who have failed with NG (Nab-paclitaxel + gemcitabine) regimen after treatment with Donafenib plus S-1.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No